CLINICAL TRIAL: NCT00951561
Title: A Randomized Four-Way Crossover Comparison Study of Pain Relief From Dysmenorrhea Between the Vipon Tampon and Ibuprofen
Brief Title: A Comparison Study of Pain Relief From Dysmenorrhea Between the Vipon Tampon and Ibuprofen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Another Way Products (Industry)
Responsible Party: Charles Tepper, Director, Another Way Products, LLC
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AWP01-01; NCT00456079 (obsolete NCT alias); NCT00587782 (obsolete NCT alias)
Record Dates: First submitted 2009-07-31; First posted 2009-08-04 (Estimated); Results first posted 2010-10-04 (Estimated); Last update posted 2011-06-16 (Estimated); Status verified 2011-06

CONDITIONS: Dysmenorrhea
Keywords: Dysmenorrhea
MeSH Terms: conditions — Dysmenorrhea | interventions — Ibuprofen; Anti-Inflammatory Agents, Non-Steroidal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vipon (Experimental)
  Interventions: Device: Vipon
- Ibuprofen (Active Comparator)
  Interventions: Drug: Ibuprofen

INTERVENTIONS:
Device: Vipon — The Vipon is a tampon with a small motor unit within, which produces vibratory stimulation, used during menstruation to provide pain relief for women with dysmenorrhea.
  Other Names: Vipon, vibrating tampon
  Arms: Vipon
Drug: Ibuprofen — 400 mg daily
  Other Names: Ibuprofen, NSAIDs
  Arms: Ibuprofen

SUMMARY:
The purpose of this study is to compare the Vipon tampon with ibuprofen in relieving pain in women with dysmenorrhea. Subjects completed a total of 4 treatment intervals; each subject was randomized to use the VIPON as their treatment for two intervals and Ibuprofen as their treatment for two intervals.

DETAILED DESCRIPTION:
Pain caused by dysmenorrhea can range from mild to severe. At least 50% of all menstruating women experience appreciable pain at some time during their menstruation. An estimated 600 million work hours are lost annually to this affliction with an average loss of time of two or more workdays per year per female employee. Treatment of dysmenorrhea may include either non-pharmacological or pharmacological measures. Pharmacological treatments include oral contraceptives to treat hormonal imbalances, over-the-counter analgesics or non-steroidal anti-inflammatory drugs. The Vipon is a tampon with a small motor unit within, which produces vibratory stimulation. This study aims to provide information on the safety and efficacy of the Vipon in a randomized controlled clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Females ages >= 18 years
* 4 consecutive monthly menstrual cycles
* Self-assessment of dysmenorrhea
* Non-pregnant status
* Agrees to use adequate birth control during the trial
* Consents to use tampons through the test of cure assessment
* Provides informed consent for participating in the trial

Exclusion Criteria:

* Prohibited use of pain medication 4 hours prior to treatment and during the first 2 hours after treatment with study medication
* Positive pregnancy test
* Unwilling or unable to comply with protocol
* Allergic to ibuprofen

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2006-11; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Truman Medical Center, Kansas City, Missouri
  - University of Kansas Medical Center, Department of Obstetrics and Gynecology, Kansas City, Missouri

RESULTS

PARTICIPANT FLOW:
Groups:
- Vipon/Ibuprofen/Vipon/Ibuprofen: Subjects participated for a total of 4 menstrual cycles. Subjects used either VIPON as a medical device or up to 2 ibuprofen tablets (each tablet containing 200 mg ibuprofen) during the first menstrual cycle. Subjects used crossover treatment during second menstrual cycle, randomized for cycle 3, and crossed over for cycle 4. All subjects used tampons for absorption of menstrual fluid during treatment and at least 2 hours post treatment. Subjects taking ibuprofen also used a tampon during treatment.
Period: Overall Study
Arm/Group | Vipon/Ibuprofen/Vipon/Ibuprofen | Ibuprofen/Vipon/Ibuprofen/Vipon | Vipon/Ibuprofen/Ibuprofen/Vipon | Ibuprofen/Vipon/Vipon/Ibuprofen
Started | 25 (Randomized Vipon or Ibuprofen period 1, crossover period 2, randomized period 3, crossover period 4) | 29 | 21 (1 subject used Vipon periods 1 & 2 instead of Ibuprofen period 2.) | 27
Completed | 25 | 29 | 18 (3 subjects dropped after period 2) | 26 (1 subject dropped after period 2)
Not Completed | 0 | 0 | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Study Participants: Subjects completed a total of 4 treatment intervals; each subject was randomized to use the VIPON as their treatment for two intervals and Ibuprofen as their treatment for two intervals.
Arm/Group | Study Participants
Number analyzed (Participants) | 102
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 102
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 32.1 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 102
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 102

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Intervention Uses That Resulted in at Least 1 Point Decrease in Pain and Requiring no Rescue Medication Using the Modified Melzack-McGill Scale Using a Mixed Model
Description: Modified Melzack-McGill Scale measures general pain (0=none, 1-3=mild, 4-6=moderate, 7-9=severe, 10=worst pain) Total Number of Uses Analyzed is a sum of the Number of Uses collected at each time point.
Time Frame: 1 month, 2 months, 3 months, 4 months
Population: Statistical analysis was carried out per plan.
Measure: Number; unit: percentage of uses
Units Other Than Participants: uses of intervention
Groups:
- VIPON; Ibuprofen: Subjects completed 4 treatment intervals; each subject was randomized to use the VIPON as their treatment during two intervals and Ibuprofen as their treatment during two intervals.
Arm/Group | VIPON | Ibuprofen
Number analyzed (Participants) | 98 | 98
Number analyzed (uses of intervention) | 191 | 192
percentage of uses | 73.8 | 75.5
Statistical Analysis 1: Comparison: VIPON vs Ibuprofen; Test type: Non-Inferiority or Equivalence — The sample size calculation is performed in nQuery version 5.0 with the following stipulations: alpha is 0.05; response for both ibuprofen and Vipon is 85%; delta is 10%; no difference in response rates is expected between the two treatment arms, and power is 80%. This calculation is performed for an equivalence/non-inferiority primary analysis; p < 0.05, Mixed Models Analysis; Difference in % of Uses from Mixed Model = -1.6

ADVERSE EVENTS:
Description: No Serious Adverse Events were deemed to be related to the VIPON.
Arm/Group | Study Participants
Serious Adverse Events (participants affected / at risk) | 2/102
Other Adverse Events (participants affected / at risk) | 48/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Participants (N=102)
Pregnancy (Reproductive system and breast disorders) | 1 (1)
Appendicitis (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Participants (N=102)
Acne (Skin and subcutaneous tissue disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (2)
Back ache (Musculoskeletal and connective tissue disorders) | 2 (2)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Cellulitis (Infections and infestations) | 1 (2)
Chest congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Cold (General disorders) | 1 (1)
Colposcopy (Reproductive system and breast disorders) | 1 (1)
Cough (General disorders) | 1 (1)
Cramps (Reproductive system and breast disorders) | 2 (2)
Cryptosporidiosis (Infections and infestations) | 1 (1)
Daytime hypersomnia (General disorders) | 1 (1)
Decreased appetite (General disorders) | 1 (1)
Dental abscess (General disorders) | 1 (1)
Dental infection (Infections and infestations) | 1 (1)
Dental pain (General disorders) | 2 (2)
Depression (Psychiatric disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Elevated blood pressure (Cardiac disorders) | 2 (2)
Fatigue (General disorders) | 1 (1)
Generalized body aches (General disorders) | 1 (1)
Giardia (Infections and infestations) | 1 (1)
Headache (General disorders) | 10 (15) — A single device-related adverse event, headache, occurred during the study and the relationship to the device was deemed "possible".
Hypercholesterolemia (General disorders) | 1 (1)
Hypertension (Cardiac disorders) | 1 (1)
Insect bite (General disorders) | 1 (2)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1)
Lymphedema (Immune system disorders) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 1 (1)
Mountain sickness (General disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Pericarditis (Cardiac disorders) | 1 (1)
Peridontal surgery (Surgical and medical procedures) | 1 (1)
Poison ivy reaction (Infections and infestations) | 1 (1)
Rash (Infections and infestations) | 1 (1)
Rectal bleeding (Gastrointestinal disorders) | 1 (1)
Respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Achilles tendon pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Ankle pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Knee pain (Musculoskeletal and connective tissue disorders) | 2 (4)
Labial biopsy (Surgical and medical procedures) | 1 (1)
Root canal (General disorders) | 1 (1)
Cyst (Infections and infestations) | 1 (1)
Shoulder pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Sinus infection (Infections and infestations) | 6 (8)
Stomach flu (General disorders) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 1 (1)
Strep throat (Infections and infestations) | 3 (3)
Sunburn (Skin and subcutaneous tissue disorders) | 1 (1)
Swollen bruised right eye (General disorders) | 1 (1)
Tick bite (General disorders) | 1 (2)
Twisted back (Musculoskeletal and connective tissue disorders) | 1 (1)
Upper respiratory infection (Infections and infestations) | 7 (7)
Urinary tract infection (Infections and infestations) | 1 (1)
Vaginal yeast infection (Infections and infestations) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI agrees not to originate or use the name of Another Way Products, LLC and/or VIPON, or any of its employees, in any publicity, news release or other public announcement, written or oral, whether to the public, press or otherwise, relating to this protocol, to any amendment herto, or to the performance here under, without the prior written consent of Another Way Products, LLC